CLINICAL TRIAL: NCT03328988
Title: Comparing Two Different Analgesic Block Methods for Postoperative Pain and Recovery After Surgery -Quadratus Lumborum Block (QLB): the Effect on Peri- and Postoperative Pain and Recovery After Radical Cystectomy
Brief Title: QLB and Radical Cystectomy, Postoperative Pain
Acronym: BladderQLB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R17008
Record Dates: First submitted 2017-05-05; First posted 2017-11-01 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Postoperative Pain; Chronic Pain Post-Proceduraal; Nausea and Vomiting, Postoperative
Keywords: bladder cancer; radical cystectomy; epidural analgesia; quadratus lumborum block; postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled study
Masking Description: Patients are randomized and allocated in blocks of ten to either epidural of QLB group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus lumborum block (Experimental): Single shot bilateral QLB, ropivacaine 75 mg (20 mL) per side, placed under ultrasound control, at the end of surgery. 22 patients will be allocated in this group.
  Interventions: Procedure: QLB
- Epidural (No Intervention): Epidural catheter (placed before anesthesia induction), ropivacaine 75 mg in 50 mL isotonic saline (1,5 mg/mL), induction bolus after surgery 1 mL/10 kg ideal weight and there on continuous infusion 2-8 mL/h according to analgesic need. 22 patients will be allocated in this group.
  This is the current standard for postoperative pain relief in cystectomy patients in our hospital

INTERVENTIONS:
Procedure: QLB — bilateral single shot block, placed under ultrasound control between the thoracolumbar fascial structures close to the quadratus lumborum muscle
  Other Names: quadratus lumborum block
  Arms: Quadratus lumborum block

SUMMARY:
There are ca 1000 new cases of bladder cancer in Finland/year. The curative therapy for high risk bladder cancer is radical cystectomy. The golden standard is still an open surgery despite development of laparoscopic techniques. Epidural analgesia is considered as most effective for the treatment of postoperative pain. However, there is a need for other effective options, because epidural analgesia has some contraindications and risks for serious complications. Recently quadratus lumborum block has gained popularity in the treatment of postoperative pain after various surgeries in the area from hip to mamilla. It is more beneficial than other peripheral blocks, since it covers also the visceral nerves. Contrary to the need of epidural catether a single shot QLB has reported to last up to 48 hours.

Inadequately treated acute postoperative pain is considered as one of the main risk factors for persistent postoperative pain.

44 patients aging 18-85 will be recruited based on a power calculation. The primary outcome measure is the acute postoperative need for rescue analgesics. Secondary outcomes are acute pain (NRS scale), nausea, vomiting, mobilisation and longterm outcomes such as quality of life and persistent pain.

DETAILED DESCRIPTION:
44 patients, uindergoing radical cystectomy, aging 18-85 will be recruited based on a power calculation. The 44 patients will be divided in 2 groups, the intervention group receiving a quadratus lumborum block (75mg ropivacaine) and the no intervention group receiving the current standard care of our hospital -an epidural.

The primary outcome measure is the acute postoperative need for rescue analgesics. Secondary outcomes are acute pain (NRS scale), nausea, vomiting, mobilisation and longterm outcomes such as quality of life and persistent pain.

ELIGIBILITY:
Inclusion Criteria:

* patients with bladder cancer coming to the open radical cystectomy.

Exclusion Criteria:

* age under 18y or over 85y,
* diabetes type 1 with complications,
* no co-operation or inadequate finnish language,
* persistent pain for other reason.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
opiate consumption | 24 hours
  intravenous patient controlled analgesia

SECONDARY OUTCOMES:
pain score | 7 days
  numerical rating scale
postoperative nausea and vomiting | 72 hours
  numerical rating scale and amount of vomites
mobilisation | 72 hours after surgery
  standing up and mobilizing
quality of life | 12 months
  SF 36
persistent pain | 12 months
  paindetect McGill
functional query | 12 months
  assessment how pain in operation region limits daily functions

CONTACTS AND LOCATIONS:
Overall Officials: Maija-Liisa Kalliomaki, PhD, Study Director — Tampere University Hospital, Department of anesthesia
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Finnish Cancer Registry. Cancer in Finland 2007-2011. Cancer Society of Finland Publication, Helsinki. 2. Witjes AJ, Lebret T, Comperat EM et al. Eur Urol. 2016 Jun 30 . 3. Azhar RA, Bochner B, Catto J et al. Eur Urol. 2016; 70: 176-187. 4. Voldby AW, Brandstrup B. Journal of Intensive Care 2016; 4:27. 5. Rawal N. Eur J Anae sthesiol 2016; 33:160 - 171 6. Kehlet H, Jensen TS, Woolf CJ . Lancet. 2006 May 13;367(9522):1618- 25 7. Gordon DB, de Leon-Casasola OA, Wu CL, ET AL. The Journal of Pain 2016; 17(2): 158-166. 8. Chou R, Gordon DB, de Leon-Casasola OA, ET AL. The Journal of Pain 2016;17(2):131-157 9. Gustavsson A., Bjorkman J., Ljungcrantz C., ET AL. Eur J Pain 2012:16 ; 289 - 299 10. Breivik H, Bang U, Jalonen J, ET AL Acta Anesthesiol Scand 20 10; 54: 16- 41. 11. Davies RG, Myles PS, Graham JM Br J Anaesth. 2006 Apr;96(4):418-26. 13. 12. Murouchi T, Iwasaki S, Yamakage M. Reg Anesth Pain Med. 2016;41:146 - 150. 13. Carney J, Finnerty O, Rauf J, ET AL. Anaesthesia. 2011;66:1023 - 30. 14. Blanco R, Ansari T, Riad W, Shetty N. Reg Anest Pain Med: Nov/Dec 2016 - vol 41 - p 757- 767. 15. Kenneth F Schulz, , Douglas G Altman, David Moher, BMJ 2010;340:c332 16. http://www.consort-statement.org
- [Derived] Veskimae E, Korgvee A, Huhtala H, Koskinen H, Kalliomaki ML, Tammela T, Junttila E. Quadratus lumborum block is feasible alternative to epidural block for postoperative analgesia after open radical cystectomy: surgical and oncological outcomes of a randomised clinical trial. Scand J Urol. 2025 Mar 13;60:59-65. doi: 10.2340/sju.v60.43105. PMID 40079670
- [Derived] Korgvee A, Veskimae E, Huhtala H, Koskinen H, Tammela T, Junttila E, Kalliomaki ML. Posterior quadratus lumborum block versus epidural analgesia for postoperative pain management after open radical cystectomy: A randomized clinical trial. Acta Anaesthesiol Scand. 2023 Mar;67(3):347-355. doi: 10.1111/aas.14188. Epub 2023 Jan 3. PMID 36547262